CLINICAL TRIAL: NCT04565223
Title: Asessing the Feasibility and Acceptability of a Cluster Randomized Study of Cognitive Behavioral Therapy for Chronic Insomnia in a Primary Care.
Brief Title: Feasibility and Acceptability of Cognitive Behavioral Therapy for Chronic Insomnia in a Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Balearic Islands Health Service (Ibsalut) (Other)
Responsible Party: Principal Investigator, Isabel Torrens, Researcher, Balearic Islands Health Service (Ibsalut)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI14/019
Record Dates: First submitted 2020-08-28; First posted 2020-09-25 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Insomnia Chronic
Keywords: primary care; cognitive behavioral therapy; clinical trial; feasibility-pilot study
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive behavioral therapy (CBT) (Experimental): 5 sessions of Cognitive behavioral therapy for insmonia and an extra session for benzodiazepine withdrawal (if necessary).
  The CBT-i included sleep hygiene counseling, stimulus control, cognitive restructuring, relaxation techniques, and benzodiazepine therapy or withdrawal
  Interventions: Behavioral: Cognitive behavioral therapy for insomnia
- Usual care (No Intervention): Usual care from GPs or nurses

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy for insomnia — is a multicomponent intervention which focuses on cognitive and behavioral factors that contribute to sleep disorders , The CBT-i included sleep hygiene counseling, stimulus control, cognitive restructuring, relaxation techniques, and benzodiazepine therapy or withdrawal (when needed). To conduct the intervention, guidelines for GPs and nurses and graphic and written materials for patients (sleep diary, registry of behavior habits, and cognitive problems) were developed
  Arms: Cognitive behavioral therapy (CBT)

SUMMARY:
This pilot-feasibility study of a cluster parallel randomized design comparing CBT-i against usual care (UC) was performed at two primary health care centers in Majorca, Spain. Patients were included if they were 18 to 65 years-old; had diagnoses of chronic insomnia according to the Insomnia Severity Index (ISI more than 8) and had insomnia longer than 3 months; and did or did not use a hypnotic medication. 25 GPs and nurses and 32 patients were randomly allocated to two groups: The outcome of the trial was improving the quality of sleep. Other primary outcomes on feasibility and applicability of the intervention were collected through nominal groups. Description of usual care was described through previous studies. Moreover we assessed recruitment process, compliance with the intervention sessions, and patient's retention.

DETAILED DESCRIPTION:
Objectives

The primary objectives of this pilot-feasibility study were:

1. To design and adapt a brief CBT-i intervention to be provided by PCPs for the treatment of chronic insomnia in individuals who are 18 to 65 years-old.
2. To define usual care (UC) for the treatment of chronic insomnia provided by PCPs as a comparative intervention (control group).
3. To assess the training activities for the CBT-i intervention by determining GPs' and nurses' satisfaction with the content and applicability of the intervention.
4. To determine the acceptability of the intervention by GPs and nurses.
5. To assess PCPs and patient recruitment, follow-up, and adherence to the intervention The secondary objective was to assess the quality of sleep in patients after 3 months of the CBT-i.

Methods Design This pilot-feasibility study of a cluster parallel randomized design comparing CBT-I against usual care (UC) was performed from September 2014 to April 2015 at two primary health care centers of Majorca (Spain) with 56,000 registered inhabitants.

Collection of information and follow up Intervention The CBT-i intervention was developed by two family physicians (IT and CV) and two psychologists (ET and MRP-P). First, a review of the literature on the use of CBT-i was performed, with a focus on interventions applied in primary care. After the literature review, the CBT-i created by Morin [24] was adapted to our setting, in which there were fewer sessions and shorter sessions. The CBT-i included sleep hygiene counseling, stimulus control, cognitive restructuring, relaxation techniques, and benzodiazepine therapy or withdrawal (when needed). To conduct the intervention, guidelines for GPs and nurses and graphic and written materials for patients (sleep diary, registry of behavior habits, and cognitive problems) were developed.

Usual care The usual treatment for persistent insomnia in a primary care setting was previously described in two cross-sectional studies performed by general practitioners and family nurses of the Primary Care Majorca Department during 2011 and 2015

ELIGIBILITY:
Inclusion criteria:

* 18 to 65 years-old
* Diagnoses of chronic insomnia according to the Insomnia Severity Index (ISI equal or higher than 8) and had insomnia longer than 3 months;
* Did or did not use a hypnotic medication.

Exclusion criteria:

* Clinical diagnosis of secondary insomnia or another sleep disorder, such as restless legs syndrome, parasomnia, or alterations of the circadian rhythm (e.g., due to shift work)
* Use of a medication that could produce sleep alterations
* Severe psychiatric disorder; depression (HADS score ≥ 8) or diagnosis of major depression in the clinical records
* Suicide attempt
* Use of an antidepressant or anti-psychotic medication
* Alcohol or drug abuse during the last year
* Reception of another CBT-i
* Sleep apnea
* Dementia or presence of a cognitive deficit (Mini Mental State Evaluation score lower than 23)
* Neurodegenerative or oncological disease with poor prognosis
* Mental or physical incapacities that impeded participation in interviews
* Acute or chronic pain secondary to a rheumatic disease or another untreated chronic disease
* Pregnancy
* Participation in a previous clinical trial in the participating health centers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2015-04-01 (Actual); Study Completion 2015-11-01 (Actual)

PRIMARY OUTCOMES:
Acceptability of the training of PCPs | 3 months postintervention
  Satisfaction with training content and its ability to provide sufficient training measured though 2 nominal groups with a previous script

SECONDARY OUTCOMES:
Feasibility of the intervention | 3 months postintervention
  Adequacy of sessions in terms of content, duration and number, fitting in PCPs agenda and patients acceptance.
Feasibility of the study design | 3 months postintervention
  Number of patients eligible identified and included, number of PCP randomized, number of patients followed up,completion of follow up and adherence to intervention sessions.
Intervention Effectiveness: Sleep | pretreatment and 3 months postintervention
  The Pittsburgh Sleep Quality Index (PSQI) is a 19-items self reported questionnaire that assesses 7 clinical components of sleep quality. Each item is rated on 0 to 3 point scale in which 0 is equal to not in the past month and 3 is equal to 3 or more times a week, with a global score range from 0 to 21. A cut off score of 5 has shown to discriminate between good and bad sleepers.
Intervention Effectiveness:Anxiety | pretreatment and 3 months postintervention
  The Hospital Anxiety and Depression Scale (HADS) measures anxiety and depression levels in the preceding week. It is 14-item self-report scale with two 7-item anxiety or depression subscales. Each item scores from 0 to 3 point scale giving maximum subscale scores of 21. Patients with scores >10 are considered to have morbidity, between 8 and 10 as borderline cases and <8 absence of relevant

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Torrens, MD, Principal Investigator — Santa Ponça health Care Center

IPD SHARING:
Plan to Share IPD: No
Data not shared

REFERENCES:
- [Derived] Torrens I, Esteva M, Vicens C, Piza-Portell MR, Vidal-Thomas MC, Vidal-Ribas C, Lorente-Montalvo P, Torres-Solera E. Assessing the feasibility and acceptability of a cluster-randomized study of cognitive behavioral therapy for chronic insomnia in a primary care setting. BMC Fam Pract. 2021 Apr 16;22(1):77. doi: 10.1186/s12875-021-01429-5. PMID 33863276